CLINICAL TRIAL: NCT02656550
Title: Uterine Transplantation and Pregnancy Induction in Women Affected by Absolute Uterine Factor Infertility
Brief Title: Uterine Transplantation and Pregnancy Induction in Women Affected by Absolute Uterine Infertility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 015-158
Record Dates: First submitted 2016-01-12; First posted 2016-01-15 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Absolute Uterine Infertility
Keywords: Uterine Transplant; AUI; Rokitansky Syndrome
MeSH Terms: conditions — Mullerian aplasia | interventions — thymoglobulin; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Uterine Transplant (Experimental): Women will undergo uterine transplantation after IVF. Donor uterus will be from either a living donor or cadaveric.
  Interventions: Procedure: Uterine Transplant

INTERVENTIONS:
Procedure: Uterine Transplant — Transplant of a uterus from either a living donor or a deceased donor.,
  Other Names: Thymoglobulin; Mycophenolate

SUMMARY:
This study aims to investigate the treatment of absolute uterine infertility (AUI) due to congenital or surgical absence of a uterus or presence of a nonfunctioning uterus. The investigators will follow a model based on a Swedish study to enroll 20 women with functioning ovaries and successfully transplant the uterus from either a living or cadaveric donor, with the goal of live birth after transplantation.

DETAILED DESCRIPTION:
INTRODUCTION

Absolute Uterine Factor Infertility (AUI) is due to congenital or surgical absence of a uterus or presence of a nonfunctional uterus. Until 2014 the only option for women affected by Absolute Uterine Factor Infertility (AUI) was adoption or surrogate motherhood.

Primary Objective

* Successful living or deceased donor uterine transplants resulting in live birth.
* Pregnancy rate via in vitro fertilization.

BACKGROUND

In 1991 the National Transplantation Pregnancy Registry (NTPR) was established to study the outcomes of female transplant recipients. In 2010 the NTPR had collected data on 2000 pregnancy outcomes. The NTRP database includes data not just on the pregnancy but on follow-up of both parents and their offspring. The first reported case of pregnancy after transplant was reported in 1958.

In 2011 25,787 solid organ transplant recipients (kidney, liver, pancreas, small bowel, heart & lung) of which:

* 9662 were women
* 3505 were of childbearing age
* 765 were less than 17 years old and could potentially become pregnant later in life.

One of the benefits of receiving a kidney, liver, pancreas, small bowel, heart or lung transplant is the underlying disease that caused the subject to have a transplant is gone, therefore fertility returns. Pregnancy after transplant is increasingly common. This has led to an accumulation of data and knowledge on how to best manage this subject population. These pregnancies are still considered high-risk. Successful pregnancy outcomes are a result of transplant and obstetrics teams working closely together.

The American Society of Transplantation (AST) recommends for solid organs that pregnancy is allowable if there has been: no rejection within the past year, there is adequate and stable graft function, no acute infections that may impact fetal growth and well-being and maintenance immunosuppression is at stable dosing. Both the NTPR and AST advise waiting one year until after transplant before conceiving. This one year wait time is associated with better maternal and neonatal outcomes and fewer obstetric complications.Based on the long term data from the NPTR on transplant recipient's pregnancy outcomes and the relative safety of immunosuppressive medications a new area of transplant is being developed. Uterine transplant may provide an additional option for women with absolute uterine infertility (AUI).

Pre-clinical research into uterine transplant has been going on for more than a decade. There have been several studies demonstrating the feasibility of Uterine Transplantation in animals, both primates and non-primates. In the last year human trials have started in Europe.

RATIONALE

In Great Britain an estimated 12000 women of childbearing age are affected by AUI. In the US the number of women affected by AUI may be in the millions considering that 9 million women of reproductive age have had a hysterectomy.

Congenital absence of the Uterus has been reported in 1/5000 women and in 2005 over 12000 women in reproductive age,15 years to 44 years have been diagnosed with congenital absence of the Uterus.

In the US, 1000 hysterectomies are performed immediately post-partum for every 1 million births.

It is estimated that 62 million women in the United States are in the reproductive age and about 15.4% may have absolute AUI, and about 7 million women may have lost their uterus to benign causes or obstetric complications. Although the statistics may offer different interpretation it seems evident that thousands of women in the United States may be interested in considering Uterine Transplantation as their best option to have children.

Previous Subject Experience

There were two reported attempts at uterine transplantation at other institutions, one of which was able to carry two pregnancies but not at term. However, the University of Gothenburg reported the first clinical trial of Uterine Transplantation as nouvelle treatment for AUI.

In this report 9 living donors and 9 recipients underwent donor hysterectomies and recipient uterine transplantation. Seven out of the 9 had viable uteri at the time of the report with 1 recipient losing the transplanted uterus to an infection and the other one to a vascular complication. One donor suffered a surgical grade IIIb complication, an ureterovaginal fistula, and was successfully treated.

This early report was followed by a subsequent one where the 7 recipients showed regular menses and 5 out of the seven recipient suffered mild rejection episodes that were all successfully treated.

The feasibility of Uterine Transplantation as a cure to AUI was finally demonstrated by the first live birth after uterus transplantation.

The surgeries have been described by the Gothenburg University Group consist of a total abdominal hysterectomy and upper vaginectomy with preservation of the major feeding arteries and veins to the uterus of the donor and the implantation of the uterus in the pelvis of the recipient. Vascular anastomosis is achieved between the two major arteries and veins of the uterus, extending to the external iliac vessels of the recipient using transplant microvascular techniques. Finally the vaginal rim of the transplanted uterus is anastomosed to the recipient's vaginal vault.

The procedure can be performed also with a uterus obtained from a deceased donor. The hysterectomy in the deceased donor will proceed as described above. The advantage will be obtaining the vascular pedicle attached to segments of the iliac artery and vein which will make the implantation in the recipient technically easier. The preservation solution will not change and the ischemia time will be kept under 6 hours.

2. STUDY DESIGN This is a prospective study to treat absolute uterine infertility (AUI) through uterine transplantation resulting in live birth.

There will be five distinct clinical stages in the study after inclusion/exclusion met criteria & subject consented: Pre-transplant/Screening, Transplant/Recovery, embryo transfer/Pregnancy, Delivery/Explant, Follow up.

Number of Clinical Sites and Subjects This trial will be conducted at the Annette C. and Harold C. Simmons Transplant Institute, Baylor University Medical Center in Dallas, TX. A total of 10 female (biologically) subjects will receive a uterine transplant. Subjects can either receive a uterus from a living donor or a cadaveric donor. Living donors will be consented per the living donor research protocol. Uterus recovery from cadaveric donors will follow UNOS guidelines.

SUBJECT PARTICIPATION and STUDY DURATION

All subjects will be followed for a 5 year period post-transplant. Continued follow up depends upon the subject status:

* Subjects who received a uterine transplant resulting in live birth then and have the uterus removed will be followed for 12 months post explant.
* Subjects who received a uterine transplant resulting in live birth and desire another pregnancy will be followed through the second pregnancy resulting in live birth for 12 months post explant.
* Subjects who have the uterus explanted due to infection, rejection or unable to maintain pregnancy will be followed for 12 months post explant.

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed with Absolute Uterine Infertility (AUI) and intact native ovaries.
2. Women of childbearing age 20-35.
3. Human papillomarvius negative or received vaccination for human papillomarvius virus (HPV). Subjects with a history of HPV in the past must show a negative history since and test negative at screening.
4. A subject who is negative for Gonorrhea, Chlamydia and Syphilis.
5. A subject with the history of Herpes (HSV-2) with no current symptoms. Subject may require preventative maintenance per study doctor discretion.
6. Subjects have received counseling regarding infertility alternatives to uterine transplant such as adoption or surrogate pregnancy.
7. Willing to undergo in-vitro fertilization and medically cleared for in-vitro fertilization.
8. Evaluated by a fertility specialist and determined to have good ovarian reproductive potential and ability to carry fetus to term.
9. Must have the ability to fund, either through third party coverage or through other their own personal financing, any expenses associated with assisted reproduction services provided to them.
10. Meets physiological recipient criteria

Exclusion Criteria:

1. Subject with Diabetes Mellitus Type I and II by medical history or elevated hemoglobin A1c blood test.
2. Subject has known hypersensitivity to Tacrolimus, Thymoglobulin or CellCept.
3. Subject with existing hypertension, per investigator's discretion.
4. Subject who has a history of solid organ or bone marrow transplant.
5. Subject who has history of cancer in last five years.
6. Subject with a body mass index >30.
7. Subject with an active infection.
8. Subject who is seropositive for HIV, HBV, HCV
9. Subject with technical obstacles as per anatomical malformations, which pose a high surgical risk in the judgment of the investigator.
10. Subject unwilling or unable to comply with study requirements.
11. Subject unable to undergo in-vitro fertilization or not cleared for transplant.
12. Subject who has smoked within the last 12 months.
13. Subject who has alcohol or drug abuse within 12 months of screening.
14. Subject with any pre-existing clinical or medical conditions that would pose the subject at an increased risk, as per the investigator's discretion.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of successful live births after uterine transplant and IVF. | 2 years after transplant
  Full term birth by cesarean section.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brannstrom M. Uterus transplantation. Curr Opin Organ Transplant. 2015 Dec;20(6):621-8. doi: 10.1097/MOT.0000000000000246. PMID 26536423
- [Background] Brannstrom M, Johannesson L, Dahm-Kahler P, Enskog A, Molne J, Kvarnstrom N, Diaz-Garcia C, Hanafy A, Lundmark C, Marcickiewicz J, Gabel M, Groth K, Akouri R, Eklind S, Holgersson J, Tzakis A, Olausson M. First clinical uterus transplantation trial: a six-month report. Fertil Steril. 2014 May;101(5):1228-36. doi: 10.1016/j.fertnstert.2014.02.024. Epub 2014 Feb 27. PMID 24582522
- [Background] Johannesson L, Kvarnstrom N, Molne J, Dahm-Kahler P, Enskog A, Diaz-Garcia C, Olausson M, Brannstrom M. Uterus transplantation trial: 1-year outcome. Fertil Steril. 2015 Jan;103(1):199-204. doi: 10.1016/j.fertnstert.2014.09.024. Epub 2014 Oct 22. PMID 25439846
- [Background] Brannstrom M, Johannesson L, Bokstrom H, Kvarnstrom N, Molne J, Dahm-Kahler P, Enskog A, Milenkovic M, Ekberg J, Diaz-Garcia C, Gabel M, Hanafy A, Hagberg H, Olausson M, Nilsson L. Livebirth after uterus transplantation. Lancet. 2015 Feb 14;385(9968):607-616. doi: 10.1016/S0140-6736(14)61728-1. Epub 2014 Oct 6. PMID 25301505
- [Background] Louden, K. (2009). Pregnancy After Transplantation: Improving Outcomes Through Counseling, Closed Management, and Research. Nephrology Times, 2(2), 11-13
- [Background] Mann, W., Goff, B., Falk, S. et. al (2015). Radical Hysterectomy. UpToDate, 3303 (9).
- [Background] Mukherjee, S. & Shapiro, R, et. al. (2011). Transplantation and Pregnancy. Kidney, 716, 1097.
- [Derived] Johannesson L, Wood-Trageser MA, Lesniak D, Punar M, Klingman L, Naziruddin B, Askar M, Demetris AJ, Testa G. Unique Lessons From the Natural Progression of Rejection in Human Uterine Allografts. Clin Transplant. 2024 Aug;38(8):e15434. doi: 10.1111/ctr.15434. PMID 39166465
- [Derived] Testa G, McKenna GJ, Wall A, Bayer J, Gregg AR, Warren AM, Lee SHS, Martinez E, Gupta A, Gunby R, Johannesson L. Uterus Transplant in Women With Absolute Uterine-Factor Infertility. JAMA. 2024 Sep 10;332(10):817-824. doi: 10.1001/jama.2024.11679. PMID 39145955
- [Derived] Johannesson L, Humphries LA, Porrett PM, Testa G, Anderson S, Walter JR, Rush M, Ferrando CA, O'Neill K, Richards EG. Classification and treatment of vaginal strictures at the donor-recipient anastomosis after uterus transplant. Fertil Steril. 2024 Sep;122(3):525-534. doi: 10.1016/j.fertnstert.2024.04.019. Epub 2024 Apr 16. PMID 38636770
- [Derived] Walter JR, Johannesson L, Falcone T, Putnam JM, Testa G, Richards EG, O'Neill KE. In vitro fertilization practice in patients with absolute uterine factor undergoing uterus transplant in the United States. Fertil Steril. 2024 Sep;122(3):397-405. doi: 10.1016/j.fertnstert.2024.04.017. Epub 2024 Apr 15. PMID 38631504
- [Derived] Johannesson L, Testa G, Petrillo N, Gregg AR. Unique risk factors for unplanned preterm delivery in the uterus transplant recipient. Hum Reprod. 2024 Jan 5;39(1):74-82. doi: 10.1093/humrep/dead240. PMID 37994646
- [Derived] Finotti M, Testa G, Koon EC, Johannesson L. Graft Hysterectomy After Uterus Transplantation With Robotic-assisted Techniques. Transplantation. 2023 Sep 1;107(9):e236-e237. doi: 10.1097/TP.0000000000004695. Epub 2023 Aug 21. No abstract available. PMID 37606907
- [Derived] Warren AM, McMinn K, Testa G, Wall A, Saracino G, Johannesson L. Motivations and Psychological Characteristics of Nondirected Uterus Donors From The Dallas UtErus Transplant Study. Prog Transplant. 2021 Dec;31(4):385-391. doi: 10.1177/15269248211046027. Epub 2021 Oct 29. PMID 34713738
- [Derived] York JR, Testa G, Gunby RT, Putman JM, McKenna GJ, Koon EC, Bayer J, Zhang L, Gregg AR, Johannesson L. Neonatal Outcomes after Uterus Transplantation: Dallas Uterus Transplant Study. Am J Perinatol. 2023 Jan;40(1):42-50. doi: 10.1055/s-0041-1727212. Epub 2021 Apr 20. PMID 33878776
- [Derived] Putman JM, Zhang L, Gregg AR, Testa G, Johannesson L. Clinical pregnancy rates and experience with in vitro fertilization after uterus transplantation: Dallas Uterus Transplant Study. Am J Obstet Gynecol. 2021 Aug;225(2):155.e1-155.e11. doi: 10.1016/j.ajog.2021.02.037. Epub 2021 Mar 12. PMID 33716072
- [Derived] Agarwal A, Johannesson L, Findeis SK, Punar M, Askar M, Ma TW, Pinto K, Demetris AJ, Testa G. Clinicopathological Analysis of Uterine Allografts Including Proposed Scoring of Ischemia Reperfusion Injury and T-cell-mediated Rejection-Dallas UtErus Transplant Study: A Pilot Study. Transplantation. 2022 Jan 1;106(1):167-177. doi: 10.1097/TP.0000000000003633. PMID 33481553
- [Derived] Johannesson L, Testa G, Putman JM, McKenna GJ, Koon EC, York JR, Bayer J, Zhang L, Rubeo ZS, Gunby RT, Gregg AR. Twelve Live Births After Uterus Transplantation in the Dallas UtErus Transplant Study. Obstet Gynecol. 2021 Feb 1;137(2):241-249. doi: 10.1097/AOG.0000000000004244. PMID 33416285
- [Derived] Johannesson L, Koon EC, Bayer J, McKenna GJ, Wall A, Fernandez H, Martinez EJ, Gupta A, Ruiz R, Onaca N, Testa G. Dallas UtErus Transplant Study: Early Outcomes and Complications of Robot-assisted Hysterectomy for Living Uterus Donors. Transplantation. 2021 Jan 1;105(1):225-230. doi: 10.1097/TP.0000000000003211. PMID 32150040
- [Derived] Warren AM, Testa G, Anthony T, McKenna GJ, Klintmalm GB, Wallis K, Koon EC, Gunby RT Jr, Johannesson L. Live nondirected uterus donors: Psychological characteristics and motivation for donation. Am J Transplant. 2018 May;18(5):1122-1128. doi: 10.1111/ajt.14670. Epub 2018 Feb 13. PMID 29364592